CLINICAL TRIAL: NCT01114945
Title: A Prospective Study Comparing Video Laryngoscopy Devices to Direct Laryngoscopy for Tracheal Intubation of Patients Undergoing Bariatric Surgery
Brief Title: Comparative Effectiveness of Intubating Devices in the Morbidly Obese
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Roya Yumul, M.D.,PhD., Residency program director, Department of anesthesiology, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Pro00019199
Record Dates: First submitted 2010-04-23; First posted 2010-05-03 (Estimated); Results first posted 2016-03-09 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-03

CONDITIONS: Obesity
Keywords: Direct Laryngoscopy; Video-Mac; GlideScope; McGrath; Laryngoscopy; Bariatrics; Glottic view; Airway intubating devices; Tracheal intubation
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Video-Mac (Experimental): Video-Mac device used during intubation procedure
  Interventions: Device: Video-Mac
- GlideScope (Experimental): GlideScope device used during intubation procedure
  Interventions: Device: GlideScope
- McGrath (Experimental): McGrath device used during intubation procedure
  Interventions: Device: McGrath
- Direct Macintosh Laryngoscopy (Active Comparator): Direct Macintosh Laryngoscopy (DL) used during intubation procedure
  Interventions: Device: Direct Macintosh Laryngoscopy

INTERVENTIONS:
Device: McGrath — Intubation with the McGrath device
  Arms: McGrath
Device: GlideScope — Intubation with the GlideScope device
  Arms: GlideScope
Device: Direct Macintosh Laryngoscopy — Intubation with Direct Macintosh Laryngoscope
  Arms: Direct Macintosh Laryngoscopy
Device: Video-Mac — Intubation with the Video-Mac device
  Arms: Video-Mac

SUMMARY:
This prospective, randomized study will compare the effectiveness of 4 different airway intubating devices which are most commonly used.

The four different devices are as follows: McGrath video laryngoscope, GlideScope video laryngoscope, Video-Mac video laryngoscope, and Macintosh size 4 direct laryngoscope.

DETAILED DESCRIPTION:
Hypothesis: the use of a video laryngoscope will improve the glottic view compared to direct laryngoscopy, and secondarily, use of the video laryngoscope will reduce the time required to achieve successful tracheal intubation in patients undergoing bariatric surgery. (Weight loss surgery). The three types of video laryngoscopy devices include; the Verethon GlideScope, LMA McGrath and Karl-Storz Video-Mac.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a documented body mass index (BMI) of >35.
* Patients scheduled to undergo inpatient surgery procedures under general anesthesia.
* Willingness and ability to sign an informed consent document
* 18 - 80 years of age
* American Society of Anesthesiologists (ASA) Class II- III adults of either sex.

Exclusion Criteria:

* Patients who are deemed to be such a significant of an airway risk that they necessitate awake fiberoptic intubation
* Patients with a history facial abnormalities, oral-pharyngeal cancer or reconstructive surgery
* Emergency surgeries
* Pregnancy
* The inability to tolerate 0.2mg of glycopyrrolate based on tachycardia.
* Any other conditions or use of any medication which may interfere with the conduct of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2010-05; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roya Yumul, MD, PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Obese patients (ASA II-III) undergoing bariatric surgery (e.g., laparoscopic gastric band placement, laparoscopic Roux-EN-Y gastric bypass laparoscopic) requiring orotracheal intubation were randomly assigned to one of four study groups.
  Enrollment from May 2010 to February 2012.
Groups:
- Video-Mac: Video-Mac device
- GlideScope: GlideScope device
- McGrath: MacGrath
- Direct Macintosh Laryngoscopy: Direct Macintosh Laryngoscopy (DL)
Period: Overall Study
Arm/Group | Video-Mac | GlideScope | McGrath | Direct Macintosh Laryngoscopy
Started | 30 | 30 | 30 | 31
Completed | 30 | 30 | 30 | 31
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Obese patients (ASA II-III). In the Direct Macintosh group there is one more participant included, this is due that the last participant declined to complete with the last assessment.
  Later changed his mind and completed the study (In that time we had enrolled another subject so we decided to use the data of both participants.
Groups:
- Direct Macintosh Laryngoscopy: Direct Macintosh Laryngoscope device
- McGrath: MacGrath device
- Total: Total of all reporting groups
Arm/Group | Direct Macintosh Laryngoscopy | Video-Mac | GlideScope | McGrath | Total
Number analyzed (Participants) | 31 | 30 | 30 | 30 | 121
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46 (12) | 44 (12) | 45 (12) | 45 (12) | 45 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 23 | 20 | 89
  Male | 8 | 7 | 7 | 10 | 32
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 42 (5) | 43 (8) | 43 (5) | 41 (6) | 42 (6)

OUTCOME MEASURES:

1. Primary Outcome: Intubation Time Using a Stop Watch
Description: Evaluate if the time it takes to achieve successful tracheal intubation in patients undergoing bariatric surgery (weight loss surgery) will be reduced using the video-mac, glidescope, and McGrath vs direct laryngoscopy.
Time Frame: up to 3 minutes
Population: Times following initial insertion of laryngoscope blade:
  to obtain glottic view (sec) to placement of tracheal tube (sec) to confirm with CO2 waveform (sec)
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Direct Macintosh Laryngoscopy | Video-Mac | GlideScope | McGrath
Number analyzed (Participants) | 31 | 30 | 30 | 30
Seconds
  Time to placement of tracheal tube | 43 (44) | 22 (15) | 45 (32) | 40 (32)
  Time to confirm with CO2 waveform | 70 (43) | 49 (25) | 69 (34) | 62 (31)

2. Primary Outcome: Time to Obtain Glottis Visualization (Seconds)
Description: It is the time (seconds) following initial insertion of laryngoscope blade to obtain a glottic view.
  Start of intubation procedure to Glottic view (the opening between the vocal cords at the upper part of the larynx) visualization comparison between the four devices in patients undergoing bariatric surgery
Time Frame: up to 1 minute
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Direct Macintosh Laryngoscopy | Video-Mac | GlideScope | McGrath
Number analyzed (Participants) | 31 | 30 | 30 | 30
Seconds | 20 (28) | 9 (8) | 12 (9) | 10 (9)

3. Primary Outcome: Percentage of Glottic Opening (POGO) [%]
Description: POGO score of 100% denotes visualization of the entire glottic opening in linear fashion from the anterior commissure to the posterior cartilages. If none of the glottic opening is seen, then the POGO score is 0%.
  View of the glottic opening (0-100%) during the intubation process.
Time Frame: up to 1 minute
Measure: Mean (Standard Deviation); unit: percentage of glottis opening
Arm/Group | Direct Macintosh Laryngoscopy | Video-Mac | GlideScope | McGrath
Number analyzed (Participants) | 31 | 30 | 30 | 30
percentage of glottis opening | 57 (41) | 84 (20) | 87 (16) | 91 (11)

4. Primary Outcome: Glottis View Using the Cormack Lehane Score
Description: Cormack Lehane score classification:
  Grade 1: Most of the glottis is visible Grade 2: At best almost half of the glottis is seen, at worst only the posterior tip of the arytenoids is seen Grade 3: Only the epiglottis is visible Grade 4: No laryngeal structures are visible
Time Frame: Up to 1 minute
Population: Cormack Lehane score (grade:1/2/3/4 [n])
Measure: Number; unit: participants
Arm/Group | Direct Macintosh Laryngoscopy | Video-Mac | GlideScope | McGrath
Number analyzed (Participants) | 31 | 30 | 30 | 30
participants
  Grade 1 | 12 | 16 | 18 | 23
  Grade 2 | 8 | 12 | 10 | 7
  Grade 3 | 5 | 2 | 2 | 0
  Grade 4 | 6 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 day
Groups:
- Video-Mac: Video-Mac device used during intubation procedure
  McGrath: McGrath will be compared with:
  Direct Macintosh Laryngoscopy Video-Mac GlideScope
  GlideScope: GlideScope will be compared with:
  Direct Macintosh Laryngoscopy Video-Mac and McGrath
  Direct Macintosh Laryngoscopy: Direct Macintosh Laryngoscopy will be compared with:
  GlideScope Video-Mac and McGrath
- GlideScope: GlideScope device used during intubation procedure
  McGrath: McGrath will be compared with:
  Direct Macintosh Laryngoscopy Video-Mac GlideScope
  Direct Macintosh Laryngoscopy: Direct Macintosh Laryngoscopy will be compared with:
  GlideScope Video-Mac and McGrath
  Video-Mac: Video-Mac will be compared with:
  Direct Macintosh Laryngoscopy GlideScope and McGrath
- McGrath: McGrath device used during intubation procedure
  GlideScope: GlideScope will be compared with:
  Direct Macintosh Laryngoscopy Video-Mac and McGrath
  Direct Macintosh Laryngoscopy: Direct Macintosh Laryngoscopy will be compared with:
  GlideScope Video-Mac and McGrath
  Video-Mac: Video-Mac will be compared with:
  Direct Macintosh Laryngoscopy GlideScope and McGrath
- Direct Macintosh Laryngoscopy: Direct Macintosh Laryngoscopy (DL) used during intubation procedure
  McGrath: McGrath will be compared with:
  Direct Macintosh Laryngoscopy Video-Mac GlideScope
  GlideScope: GlideScope will be compared with:
  Direct Macintosh Laryngoscopy Video-Mac and McGrath
  Video-Mac: Video-Mac will be compared with:
  Direct Macintosh Laryngoscopy GlideScope and McGrath
Arm/Group | Video-Mac | GlideScope | McGrath | Direct Macintosh Laryngoscopy
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 0/31
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No